CLINICAL TRIAL: NCT07291609
Title: Microplastics and Nanoplastics in Patients With Chronic Coronary Syndromes
Acronym: CCS-Plastics
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliera "Sant'Andrea" (Other)
Collaborators: University of Campania Luigi Vanvitelli (Other); Azienda Ospedaliera Universitaria Integrata Verona (Other); Morgagni Pierantoni Hospital (Other); Azienda Ospedaliera Sant'Anna e San Sebastiano (Other); Centro Cardiologico Monzino, Milan, Italy (Unknown)
Responsible Party: Principal Investigator, Emanuele Barbato, Full Professor, Azienda Ospedaliera "Sant'Andrea"
Other Study IDs: 1000/2025
Record Dates: First submitted 2025-11-24; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Chronic Coronary Syndrome; Microplastics; Nanoplastics; Coronary Artery Disease; Coronary Plaque; Computed Tomography; Pollution Exposure
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CCS patients with presence of micro- and nano-plastics (MNPs+): Consecutive patients undergoing coronary CT angiography (CCTA) for suspected or known chronic coronary syndromes (CCS) referred to invasive coronary angiography for clinical indication with the presence of micro- and nano-plastics (MNPs +).
- CCS patients without the presence of micro- and nano-plastics (MNPs-): Consecutive patients undergoing coronary CT angiography (CCTA) for suspected or known chronic coronary syndromes (CCS) referred to invasive coronary angiography for clinical indication without the presence of micro- and nano-plastics (MNPs -).

SUMMARY:
The CCS-plastics is an investigator-initiated, prospective, multicenter study of patients undergoing coronary CT angiography (CCTA) for suspected or known chronic coronary syndromes (CCS) referred to invasive coronary angiography for clinical indication. Patients identified as eligible for the protocol will be asked for written consent to participate in the study. The patients' dossiers will be uploaded and transmitted to the core laboratory for analysis. The routine management of the CCS patients will not be affected and all patients will be managed according to current standards. Invasive coronary angiography and coronary blood samples will be performed following the current standards, guidelines, and indications. During invasive coronary angiography, coronary blood samples will be collected per standard of care and sent to a centralized, specialized core laboratory for MNPs and biomarkers analysis. The central core lab for MNPs analyses will be the University of Campania Luigi Vanvitelli, Naples, Italy. The identification, quantification (concentration, mcg/ml), and typing of plastic particles will be performed in each tube for each patient, using pyrolysis-gas chromatography-mass spectrometry (Py-GC/MS) and laser direct infrared (LDIR) spectroscopy. The CCTA will be centrally analyzed by Centro Cardiologico Monzino to evaluate qualitative and quantitative plaque features. Patients will be followed clinically at 1 and 3 years per standard of care.

ELIGIBILITY:
Inclusion Criteria:

ALL the following:

1. Age > 18 years old;
2. Suspected or known chronic coronary syndromes undergoing coronary CT angiography;
3. Clinical indication to invasive coronary angiography;
4. Able to give informed consent.

Exclusion Criteria:

1. Coronary CT angiography not available;
2. Poor quality CCTA;
3. Absence of native coronary stenosis >=50% at CCTA;
4. Contraindications to invasive coronary angiography and percutaneous coronary intervention
5. Life expectancy < 1 year due to non-cardiac pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing coronary CT angiography (CCTA) for suspected or known chronic coronary syndromes (CCS) referred to invasive coronary angiography for clinical indication.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Burden of micro- and nanoplastics (MNPs) in the coronary blood of patients with chronic coronary syndromes (CCS) and obstructive coronary artery disease (CAD) | From enrollment until the date of hospital discharge, assessed up to 7 days
  To measure the burden (concentration, mcg/ml) of micro- and nanoplastics (MNPs) in the coronary blood of patients with chronic coronary syndromes (CCS) and obstructive CAD (diameter stenosis>50%)
Burden of micro- and nanoplastics (MNPs) in the coronary blood of patients with chronic coronary syndromes (CCS) and plaque features at coronary computed tomography angiography. | From enrollment until the date of hospital discharge, assessed up to 7 days
  Correlation of the burden (concentration, mcg/ml) of micro- and nanoplastics (MNPs) in the coronary blood of patients with chronic coronary syndromes (CCS) with quantitative and qualitative plaque features at coronary computed tomography angiography.

SECONDARY OUTCOMES:
Correlation of the burden of micro- and nanoplastics (MNPs) in the coronary blood of patients with chronic coronary syndromes (CCS) with diameter stenosis at coronary computed tomography angiography (CCTA). | From enrollment until the date of hospital discharge, assessed up to 7 days.
  To correlate the burden (concentration, mcg/ml) of micro- and nanoplastics (MNPs) in the coronary blood of patients with chronic coronary syndromes (CCS) with the diameter stenosis at coronary computed tomography angiography (CCTA).
Correlation of the burden of micro- and nanoplastics (MNPs) in the coronary blood of patients with chronic coronary syndromes (CCS) with plaque burden at coronary computed tomography angiography (CCTA). | From enrollment until the date of hospital discharge, assessed up to 7 days
  To correlate the burden (concentration, mcg/ml) of micro- and nanoplastics (MNPs) in the coronary blood of patients with chronic coronary syndromes (CCS) with plaque burden at coronary computed tomography angiography (CCTA).
Correlation of the burden of micro- and nanoplastics (MNPs) in the coronary blood of patients with chronic coronary syndromes (CCS) with plaque morphology at coronary computed tomography angiography (CCTA). | From enrollment until the date of hospital discharge, assessed up to 7 days
  To correlate the burden (concentration, mcg/ml) of micro- and nanoplastics (MNPs) in the coronary blood of patients with chronic coronary syndromes (CCS) with plaque morphology at coronary computed tomography angiography (CCTA).
Correlation of the burden of micro- and nanoplastics (MNPs) in the coronary blood of patients with chronic coronary syndromes (CCS) with the presence of high-risk plaque features at coronary computed tomography angiography (CCTA). | From enrollment until the date of hospital discharge, assessed up to 7 days
  To correlate the burden (concentration, mcg/ml) of micro- and nanoplastics (MNPs) in the coronary blood of patients with chronic coronary syndromes (CCS) with the presence of high-risk plaque features at coronary computed tomography angiography (CCTA).
Correlation of the burden of micro- and nanoplastics (MNPs) in the coronary blood of patients with chronic coronary syndromes (CCS) with the presence and burden of calcium at coronary computed tomography angiography (CCTA). | From enrollment until the date of hospital discharge, assessed up to 7 days.
  To correlate the burden (concentration, mcg/ml) of micro- and nanoplastics (MNPs) in the coronary blood of patients with chronic coronary syndromes (CCS) with the presence and burden of calcium at coronary computed tomography angiography (CCTA).
Correlation of the burden of micro- and nanoplastics (MNPs) in the coronary blood of patients with chronic coronary syndromes (CCS) with the pericoronary fat attenuation index at coronary computed tomography angiography (CCTA). | From enrollment until the date of hospital discharge, assessed up to 7 days
  To correlate the burden (concentration, mcg/ml) of micro- and nanoplastics (MNPs) in the coronary blood of patients with chronic coronary syndromes (CCS) with the pericoronary fat attenuation index at coronary computed tomography angiography (CCTA).
Correlation of the burden of micro- and nanoplastics (MNPs) in patients with chronic coronary syndromes (CCS) with vessel-specific ischemia. | From enrollment until the date of hospital discharge, assessed up to 7 days
  To correlate the burden (concentration, mcg/ml) of micro- and nanoplastics (MNPs) in patients with chronic coronary syndromes (CCS) with vessel-specific ischemia.
Correlation of the burden of micro- and nanoplastics (MNPs) in patients with chronic coronary syndromes (CCS) with platelet reactivity | From enrollment until the date of hospital discharge, assessed up to 7 days
  To correlate the burden (concentration, mcg/ml) of micro- and nanoplastics (MNPs) in patients with chronic coronary syndromes (CCS) with platelet reactivity as assessed by aggregometry.
Correlation of the burden of micro- and nanoplastics (MNPs) in patients with chronic coronary syndromes (CCS) with the occurrence of periprocedural events. | From enrollment until the date of hospital discharge, assessed up to 7 days
  To correlate the burden (concentration, mcg/ml) of micro- and nanoplastics (MNPs) in patients with chronic coronary syndromes (CCS) with the occurrence of periprocedural events.
Correlation of the burden of micro- and nanoplastics (MNPs) with major adverse cardiovascular events (cardiovascular death, myocardial infarction, any revascularization, hospitalization for heart failure) at 1-year follow-up. | From enrollment to 1-year follow-up.
  To correlate the burden (concentration, mcg/ml) of micro- and nanoplastics (MNPs) in patients with chronic coronary syndromes (CCS) with major adverse cardiovascular events (cardiovascular death, myocardial infarction, any revascularization, hospitalization for heart failure) at 1-year follow-up.
Correlation of the burden of micro- and nanoplastics (MNPs) in patients with chronic coronary syndromes (CCS) with all-cause death at 1-year follow-up. | From enrollment to 1-year follow-up.
  To correlate the burden (concentration, mcg/ml) of micro- and nanoplastics (MNPs) in patients with chronic coronary syndromes (CCS) with all-cause death at 1-year follow-up.
Correlation of the burden of micro- and nanoplastics (MNPs) in patients with chronic coronary syndromes (CCS) with cardiovascular death at 1-year follow-up. | From enrollment to 1-year follow-up.
  To correlate the burden (concentration, mcg/ml) of micro- and nanoplastics (MNPs) in patients with chronic coronary syndromes (CCS) with cardiovascular death at 1-year follow-up.
The correlation of the burden of micro- and nanoplastics (MNPs) in patients with chronic coronary syndromes (CCS) with myocardial infarction at 1-year follow-up. | From enrollment to 1-year follow-up.
  To correlate the burden (concentration, mcg/ml) of micro- and nanoplastics (MNPs) in patients with chronic coronary syndromes (CCS) with myocardial infarction at 1-year follow-up.
The correlation of the burden of micro- and nanoplastics (MNPs) in patients with chronic coronary syndromes (CCS) with any revascularization at 1-year follow-up. | From enrollment to 1-year follow-up.
  To correlate the burden (concentration, mcg/ml) of micro- and nanoplastics (MNPs) in patients with chronic coronary syndromes (CCS) with any revascularization at 1-year follow-up.
Correlation of the burden of micro- and nanoplastics (MNPs) in patients with chronic coronary syndromes (CCS) with hospitalization for heart failure at 1-year follow-up. | From enrollment to 1-year follow-up.
  To correlate the burden (concentration, mcg/ml) of micro- and nanoplastics (MNPs) in patients with chronic coronary syndromes (CCS) with hospitalization for heart failure at 1-year follow-up.
Correlation of the burden of micro- and nanoplastics (MNPs) with major adverse cardiovascular events (cardiovascular death, myocardial infarction, any revascularization, hospitalization for heart failure) at 3-year follow-up. | From enrollment to 3-year follow-up.
  To correlate the burden (concentration, mcg/ml) of micro- and nanoplastics (MNPs) in patients with chronic coronary syndromes (CCS) with major adverse cardiovascular events (cardiovascular death, myocardial infarction, any revascularization, hospitalization for heart failure) at 3-year follow-up.
Correlation of the burden of micro- and nanoplastics (MNPs) in patients with chronic coronary syndromes (CCS) with all-cause death at 3-year follow-up. | From enrollment to 3-year follow-up.
  To correlate the burden (concentration, mcg/ml) of micro- and nanoplastics (MNPs) in patients with chronic coronary syndromes (CCS) with all-cause death at 3-year follow-up.
Correlation of the burden of micro- and nanoplastics (MNPs) in patients with chronic coronary syndromes (CCS) with cardiovascular death at 3-year follow-up. | From enrollment to 3-year follow-up.
  To correlate the burden (concentration, mcg/ml) of micro- and nanoplastics (MNPs) in patients with chronic coronary syndromes (CCS) with cardiovascular death at 3-year follow-up.
Correlation of the burden of micro- and nanoplastics (MNPs) in patients with chronic coronary syndromes (CCS) with myocardial infarction at 3-year follow-up. | From enrollment to 3-year follow-up.
  To correlate the burden (concentration, mcg/ml) of micro- and nanoplastics (MNPs) in patients with chronic coronary syndromes (CCS) with myocardial infarction at 3-year follow-up.
Correlation of the burden of micro- and nanoplastics (MNPs) in patients with chronic coronary syndromes (CCS) with any revascularization at 3-year follow-up. | From enrollment to 3-year follow-up.
  To correlate the burden (concentration, mcg/ml) of micro- and nanoplastics (MNPs) in patients with chronic coronary syndromes (CCS) with any revascularization at 3-year follow-up.
Correlation of the burden of micro- and nanoplastics (MNPs) in patients with chronic coronary syndromes (CCS) with hospitalization for heart failure at 3-year follow-up | From enrollment to 3-year follow-up.
  To correlate the burden (concentration, mcg/ml) of micro- and nanoplastics (MNPs) in patients with chronic coronary syndromes (CCS) with hospitalization for heart failure at 3-year follow-up

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (6):
  - Division of Cardiology, A.O.R.N. "Sant'Anna e San Sebastiano", Caserta, Italy., Caserta
  - Cardiovascular Division, Morgagni-Pierantoni University Hospital, Forlì, Italy., Forlì
  - Centro Cardiologico Monzino, Milan
  - Department of Advanced Medical and Surgical Sciences, University of Campania-Luigi Vanvitelli, Naples, Italy., Napoli
  - Sant'Andrea University Hospital, Roma
  - Azienda Ospedaliera Integrata Verona, Italy, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee DH. Microplastics and Cardiovascular Diseases: Importance of Coexisting Environmental Pollutants. Circulation. 2024 Sep 17;150(12):908-910. doi: 10.1161/CIRCULATIONAHA.124.069801. Epub 2024 Sep 16. No abstract available. PMID 39283932
- [Background] Wang T, Yi Z, Liu X, Cai Y, Huang X, Fang J, Shen R, Lu W, Xiao Y, Zhuang W, Guo S. Multimodal detection and analysis of microplastics in human thrombi from multiple anatomically distinct sites. EBioMedicine. 2024 May;103:105118. doi: 10.1016/j.ebiom.2024.105118. Epub 2024 Apr 13. PMID 38614011
- [Background] Marfella R, Prattichizzo F, Sardu C, Fulgenzi G, Graciotti L, Spadoni T, D'Onofrio N, Scisciola L, La Grotta R, Frige C, Pellegrini V, Municino M, Siniscalchi M, Spinetti F, Vigliotti G, Vecchione C, Carrizzo A, Accarino G, Squillante A, Spaziano G, Mirra D, Esposito R, Altieri S, Falco G, Fenti A, Galoppo S, Canzano S, Sasso FC, Matacchione G, Olivieri F, Ferraraccio F, Panarese I, Paolisso P, Barbato E, Lubritto C, Balestrieri ML, Mauro C, Caballero AE, Rajagopalan S, Ceriello A, D'Agostino B, Iovino P, Paolisso G. Microplastics and Nanoplastics in Atheromas and Cardiovascular Events. N Engl J Med. 2024 Mar 7;390(10):900-910. doi: 10.1056/NEJMoa2309822. PMID 38446676
- [Background] Prattichizzo F, Ceriello A, Pellegrini V, La Grotta R, Graciotti L, Olivieri F, Paolisso P, D'Agostino B, Iovino P, Balestrieri ML, Rajagopalan S, Landrigan PJ, Marfella R, Paolisso G. Micro-nanoplastics and cardiovascular diseases: evidence and perspectives. Eur Heart J. 2024 Oct 7;45(38):4099-4110. doi: 10.1093/eurheartj/ehae552. PMID 39240674
- [Background] Liu S, Wang C, Yang Y, Du Z, Li L, Zhang M, Ni S, Yue Z, Yang K, Wang Y, Li X, Yang Y, Qin Y, Li J, Yang Y, Zhang M. Microplastics in three types of human arteries detected by pyrolysis-gas chromatography/mass spectrometry (Py-GC/MS). J Hazard Mater. 2024 May 5;469:133855. doi: 10.1016/j.jhazmat.2024.133855. Epub 2024 Feb 21. PMID 38428296